CLINICAL TRIAL: NCT00030849
Title: Phase II Trial Of Oral Bexarotene (Targretin) Combined With Interferon Alfa-2b (Intron-A) For Patients With Cutaneous T-Cell Lymphoma
Brief Title: Bexarotene and Interferon Alfa in Treating Patients With Cutaneous T-Cell Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000069202; MSKCC-01128; NCI-G01-2049
Record Dates: First submitted 2002-02-14; First posted 2003-01-27 (Estimated); Last update posted 2013-04-04 (Estimated); Status verified 2009-12

CONDITIONS: Lymphoma
Keywords: stage I cutaneous T-cell non-Hodgkin lymphoma; stage II cutaneous T-cell non-Hodgkin lymphoma; stage III cutaneous T-cell non-Hodgkin lymphoma; stage IV cutaneous T-cell non-Hodgkin lymphoma; recurrent cutaneous T-cell non-Hodgkin lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, T-Cell, Cutaneous | interventions — Interferon-alpha; Bexarotene

INTERVENTIONS:
Biological: recombinant interferon alfa
Drug: bexarotene

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Interferon alfa may interfere with the growth of cancer cells. Combining chemotherapy with interferon alfa may kill more cancer cells.

PURPOSE: Phase II trial to study the effectiveness of combining bexarotene with interferon alfa in treating patients who have cutaneous T-cell lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the response rate and response duration in patients with cutaneous T-cell lymphoma when treated with bexarotene and, in the absence of a complete response, interferon alfa.
* Determine the safety and toxicity in patients treated with this regimen.

OUTLINE: This is a multicenter study.

Patients receive oral bexarotene once daily for 8 weeks.

Patients with a complete response (CR) after 8 weeks continue bexarotene alone for at least another 8 weeks in the absence of unacceptable toxicity.

Patients who progress or relapse during bexarotene therapy or who achieve less than a CR after 8 weeks begin receiving interferon alfa subcutaneously 3 times a week and oral bexarotene daily for at least another 8 weeks in the absence of continuing disease progression or unacceptable toxicity.

Patients are followed at 4 weeks.

PROJECTED ACCRUAL: A total of 20-45 patients will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed cutaneous T-cell lymphoma

  * Stage IB, IIA, IIB, III, or IV
* Measurable or assessable disease

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Karnofsky 60-100%

Life expectancy:

* Not specified

Hematopoietic:

* Hemoglobin at least 9 g/dL
* WBC at least 1,500/mm^3
* Platelet count at least 70,000/mm^3

Hepatic:

* Bilirubin no greater than 2.0 mg/dL
* SGOT and SGPT no greater than 3 times upper limit of normal (ULN)
* Alkaline phosphatase no greater than 3 times ULN
* Fasting triglyceride normal (normalization with an antilipemic agent is allowed prior to study)
* No severe decompensated liver disease (e.g., cirrhosis, autoimmune hepatitis, or any other significant liver dysfunction)

Renal:

* Calcium no greater than 11.5 mg/dL
* Creatinine no greater than 2 times ULN

Cardiovascular:

* No myocardial infarction in the past 6 months
* No unstable angina
* No class III or IV congestive heart failure
* No ventricular tachyarrhythmias

Pulmonary:

* No pulmonary infiltrates or clinical pulmonary impairment

Other:

* HIV negative
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use 2 forms of effective contraception for 1 month before, during, and for 1 month after study therapy
* No known allergy or sensitivity to interferon alfa or bexarotene or other components of study drugs
* No uncontrolled thyroid disorder
* No other concurrent serious medical illness that would preclude study
* No infection
* No history of pancreatitis
* No history of neuropsychiatric disorders requiring hospitalization
* No history of autoimmune disease that would pose significant risk
* Must be willing and able to avoid prolonged exposure to the sun or ultraviolet light

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* No concurrent systemic anticancer chemotherapy

Endocrine therapy:

* No concurrent systemic corticosteroids

Radiotherapy:

* No concurrent localized radiotherapy to target lesions unless considered
* to have shown progressive disease

Surgery:

* Not specified

Other:

* At least 30 days since prior systemic doses of more than 15,000 IU per day of vitamin A or any other retinoid class drug
* At least 30 days since prior participation in any other investigational drug study
* No concurrent systemic anti-psoriatic drugs or therapies
* No concurrent systemic other anticancer drugs or therapies
* No concurrent gemfibrozil
* No other concurrent investigational medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-10; Primary Completion 2004-09 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David J. Straus, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (5):
- United States (5):
  - University of Miami Sylvester Comprehensive Cancer Center, Miami, Florida
  - NYU School of Medicine's Kaplan Comprehensive Cancer Center, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Abramson Cancer Center of the University of Pennsylvania Medical Center, Philadelphia, Pennsylvania
  - University of Texas - MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- [Result] Straus DJ, Duvic M, Kuzel T, Horwitz S, Demierre MF, Myskowski P, Steckel S. Results of a phase II trial of oral bexarotene (Targretin) combined with interferon alfa-2b (Intron-A) for patients with cutaneous T-cell lymphoma. Cancer. 2007 May 1;109(9):1799-803. doi: 10.1002/cncr.22596. PMID 17366595